CLINICAL TRIAL: NCT01651546
Title: Development and Psychometric Validation of a Scale Assessing "the Acceptance" of Clean Intermittent Self Catheterization in a Neurological and no Neurological Population With Indication to Self Catheterization.
Brief Title: Intermittent Catheterization Acceptance Test
Acronym: I-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NI11029; AOM 11014 (Other: Assistance Publique)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Intermittent Self Catheterization
Keywords: Clean Intermittent Self Catheterization; acceptance; test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Other): Patients with dysvoiding function and chronic urinary retention, with an indication to CISC.
  Interventions: Behavioral: Intermittent catheterization test

INTERVENTIONS:
Behavioral: Intermittent catheterization test — I-CAT will be a self assessment questionnaire and a simple, comprehensive and quickly passed questionnaire.

SUMMARY:
The aim of the study is to create and validate a specific test named Intermittent Catheterization Acceptance Test (I-CAT), assessing "the acceptance" of clean intermittent self catheterization (CISC) in a neurological and no neurological population with indication to self catheterization.

CISC avoids urological complications in bladder with chronic and improves quality of life. Despite theses challenges, the learning of CISC can face some physical, cognitive and psychological difficulties. Recently, we have validate a new test for predicting the physical and cognitive abilities to practice CISC named "PP-Test". Meanwhile, psychological factors are not explored in this test. To our knowledge, no study has been conducted in order to demonstrate in a prospective trial, which kind of psychological barriers can exist. Likewise it would be interesting to create a new test assessing the psychological "acceptance" of the patients to CISC before learning (I-CAT). Based on the results of this self-assessment test, the specific nurse could then change her speech by playing down the importance of some fear and anxiety described by the patients. The learning of CISC would be facilitated.

DETAILED DESCRIPTION:
The first version of the questionnaire (I-CAT) has already been elaborated from some neuro-urology experts and patients's comments.

The final version will be validated after a feasibility study. The psychometric criteria will be validated.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with neurological disease (brain, trauma and no trauma spinal injury, cauda equine syndrome) or non neurological disease
* Patients seen in consultation or in traditional hospital
* Indication for the realization of self-catheterization Intermittent must be asked because of a bladder-type retentionist or overactive bladder with an indication of medical (anticholinergics or botulinum toxin intra-detrusor injection) or surgical (kind of expansion enterocystoplasty) treatment to prevent bladder emptying without urinary catheterization
* PP-Test score ≥10/15
* Age > 18 years
* Patient with social security

Exclusion Criteria:

* Urethral injury preventing the practice of self-catheterization
* Indication to installing a suprapubic catheter or probe
* Patients able to answer to questionnaire and communicate in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intermittent catheterization acceptance test (I-CAT) | 2 years
  In order to validate the questionnaire, the patients will have to respond to I-CAT at 3 times:
  * the day the CISC's indication is decided
  * at the learning'CISC consultation about 8 days later
  * during the verification's CISC consultation about 15 days later

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PU/PH, Principal Investigator — Assistance Publique
Locations (1):
- Service Neuro-Urologie, Paris, France